CLINICAL TRIAL: NCT01455259
Title: Phase I/IIa AdCD40L Immunogene Therapy for Patients With Advanced Malignant Disease.
Brief Title: Phase I/IIa AdCD40L Immunogene Therapy for Malignant Melanoma and Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002:CD40L
Record Dates: First submitted 2011-10-11; First posted 2011-10-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Malignant Melanoma
Keywords: AdCD40L; Adenoviral vector; CD40L; CD154; malignant melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdCD40L (Experimental): Treatments once a week with 2.5x10e11 VP AdCD40L, maximum 4 treatments (total dose 1x10e12 VP). If no effect in less than 2 out of 6 melanoma patients, the following 9 melanoma patients and 6 patients with other solid tumors will receive preconditioning therapy 1-2 days prior to first and last treatment with 300mg/m2 cyclophosphamid. The next 9 melanoma patients will receive one local radiotherapy.
  Interventions: Biological: AdCD40L

INTERVENTIONS:
Biological: AdCD40L — Adenoviral serotype 5 vector, E1/E3 deleted. Human CD40L gene insert driven by RSV promoter. Vector diluted in infusion solution, 500uL solution containing 2.5x10e11 VP is intratumorally injected/treatment.

SUMMARY:
In this phase I/II trial, immunostimulatory gene therapy (AdCD40L) will be investigated. In Part 1 patients with melanoma will receive AdCD40L as mono therapy. In Part 2A, patients with melanoma and patients with other solid tumors will receive AdCD40L in combination with low dose cyclophosphamide. In Part 2B, patients with melanoma will receive AdCD40L in combination with one local radiotherapy and cyclophosphamide.

DETAILED DESCRIPTION:
In this phase I/II trial, immunostimulatory gene therapy (AdCD40L) will be investigated. In Part 1 patients with melanoma (n=6) will receive AdCD40L as mono therapy. In Part 2A, patients with melanoma (n=9) and patients with other solid tumors (n=6) will receive AdCD40L in combination with low dose cyclophosphamide. In Part 2B, patients with melanoma will receive AdCD40L in combination with one local radiotherapy and cyclophosphamide. AdCD40L is given by weekly injections of 2.5x10e11 VP, 4x; total dose 1x10e12 VP. A maximum of 30 patients will be included in this trial.

AdCD40L is an adenoviral nonreplicating vector carrying the human CD40L gene. AdCD40L infects tumor cells upon intratumoral injection and deliver the CD40L gene into the cells whereupon the virus is destroyed. CD40L is then expressed as a membrane-bound protein and interacts with the CD40 receptor expressed by for example dendritic cells (DCs) in the tumor area. DCs mature upon CD40/CD40L interactions and activates tumor-specific T cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of malignant solid cancer, ECOG 0-2.
* Disease progression on established treatments or patients not eligible to standard options.
* Signed informed consent must be obtained.

Exclusion Criteria:

* Pregnancy.
* Life expectancy less than 3 months.
* Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
* Patients with severe systemic autoimmune disease.
* Patients that do not consent to that tissue and blood samples are stored in a biobank.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
All cause adverse events | during 10 weeks
  Adverse events will be documented such as inflammation, fever, pain, changes in blood pressure, pulse etc.
Immune reactions to adenovirus and spreading of vector | during 10 weeks
  Immune reactions to adenovirus will be measured by evaluating the increase of anti-adenoviral antibodies in the patients at different time points using an ELISA. Spreading of vector will be evaluated by real time PCR to detect adenovirus vector copies in blood (plasma and erythrocyte fraction).

SECONDARY OUTCOMES:
Tumor burden as measured by PET/CT and whole body MR | At enrollment, week 5 and week 9

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Tötterman, MD, PhD, Study Chair — Uppsala University; Gustav Ullenhag, MD, PhD, Principal Investigator — Uppsala University Hospital; Angelica SI Loskog, PhD, Study Director — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Schiza A, Wenthe J, Mangsbo S, Eriksson E, Nilsson A, Totterman TH, Loskog A, Ullenhag G. Adenovirus-mediated CD40L gene transfer increases Teffector/Tregulatory cell ratio and upregulates death receptors in metastatic melanoma patients. J Transl Med. 2017 Apr 20;15(1):79. doi: 10.1186/s12967-017-1182-z. PMID 28427434